CLINICAL TRIAL: NCT03520166
Title: Treatment of Overactive Bladder, Lower Urinary Tract Symptoms and Pelvic Pain With Medium Frequency Electrotherapy (Interferential Currents)
Brief Title: Use of Medium Frequency Electrotherapy in the Treatment of OAB, LUTS and Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisioterapia Pélvica Avanzada Madrid, SRL (Other)
Responsible Party: Principal Investigator, Cristina Naranjo Ortiz, Principal Investigator, Fisioterapia Pélvica Avanzada Madrid, SRL
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPA01/2014; 1.010.817 (Other Grant/Funding Number: FUNDACION ALFONSO X)
Record Dates: First submitted 2018-04-16; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Urinary Bladder, Overactive; Lower Urinary Tract Symptoms; Pelvic Pain
Keywords: urgency; frequency; overactive bladder; LUTS; pelvic pain; electrostimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Lower Urinary Tract Symptoms; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, longitudinal, pre-/post-. Level of evidence II/III.
Masking Description: Type inclusion was consecutively type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Placebo Comparator): No treatment
  Interventions: Other: No treatment
- Group-B (Experimental): Medium frequency electrotherapy (interferential currents)
  Interventions: Other: Medium frequency electrotherapy (interferential currents)

INTERVENTIONS:
Other: Medium frequency electrotherapy (interferential currents) — Treatment with medium frequency electrotherapy, interferential currents between 5500 Hz and 8500 Hz (Combi-200®, Gymna®), was performed using transvaginal application. The frequency was increased progressively over the first six sessions (twice a week), starting with a frequency of 5500 Hz until reaching a frequency of 8500 Hz, which remained until the end of treatment.
  Arms: Group-B
Other: No treatment — No treatment
  Arms: Group-A

SUMMARY:
The aim of this study is to assess the effectiveness of medium frequency electrotherapy (interferential currents) treatment for overactive bladder (OAB), lower urinary tract symptoms (LUTS) and pelvic pain

DETAILED DESCRIPTION:
This study consists of 100 women, complaining of increased bladder sensation and urgency with or without incontinence as principal symptomatology and who had not received previous pharmacological treatment. Group-A was used as a control group (n = 50). Group-B patients received 18 sessions of medium frequency electrotherapy during 9 weeks, 2 weekly sessions

ELIGIBILITY:
Inclusion Criteria:

Increased bladder sensation Urgency Overactive bladder Lower urinary tract symptoms Pelvic pain

Exclusion Criteria:

Neurogenic bladder Acute urinary infection Pelvic floor surgery Congenital urological malformations Age less than 18 years Bladder organic pathology Pelvic radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
urgency | 24 hours
  with or without urge incontinence, usually with frequency and nocturia, can be described as the overactive bladder syndrome, urge syndrome or urgency-frequency syndrome. Measured with 24 hour voiding diary.

SECONDARY OUTCOMES:
urge urinary incontinence | 24 hours
  is the complaint of involuntary leakage accompanied by or immediately preceded by urgency. Measured with 24 hour voiding diary.
increased daytime frequency | 24 hours
  is the complaint by the patient who considers that he/she voids too often by day. Measured with 24 hour voiding diary.
nocturia | 24 hours
  is the complaint that the individual has to wake at night one or more times to void. Measured with 24 hour voiding diary.
increased bladder sensation | 24 hours
  the individual feels an early and persistent desire to void. Measured with 24 hour voiding diary.
feeling of incomplete emptying | 24 hours
  is a self-explanatory term for a feeling experienced by the individual after passing urine. Measured with 24 hour voiding diary.
nocturnal enuresis | 24 hours
  is the complaint of loss of urine occurring during sleep. Measured with 24 hour voiding diary.
incontinence | 24 hours
  is the complaint of any involuntary leakage of urine. Measured with 24 hour voiding diary.
pelvic pain | 24 hours
  is less well defined than, for example, bladder, urethral or perineal pain and is less clearly related to the micturition cycle or to bowel function and is not localised to any single pelvic organ. Measured with pain visual analogic pain scale single-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Naranjo-Ortiz, Ph.D, Principal Investigator — Fisioterapia Pelvica Avanzada Madrid, SRL

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Background] Almeida CC, Silva VZMD, Junior GC, Liebano RE, Durigan JLQ. Transcutaneous electrical nerve stimulation and interferential current demonstrate similar effects in relieving acute and chronic pain: a systematic review with meta-analysis. Braz J Phys Ther. 2018 Sep-Oct;22(5):347-354. doi: 10.1016/j.bjpt.2017.12.005. Epub 2018 Feb 2. PMID 29426587
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03520166/SAP_000.pdf
  • Study Protocol (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03520166/Prot_001.pdf